CLINICAL TRIAL: NCT02967926
Title: Digital SpyGlass Cholangioscopy Confirmed Common Bile Duct Stones Clearance Without Fluoroscopy
Brief Title: Digital SpyGlass Confirmed Common Bile Duct Stones Clearance Without Fluoroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Thanawat Luangsukrerk, Gastrointestinal Endoscopy Excellence Center, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 791/2016
Record Dates: First submitted 2016-11-03; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Common Bile Duct Diseases; Stone - Biliary; Cholangitis, Sclerosing
Keywords: common bile duct stone; cholangioscopy; SpyGlass; non-fluoroscopic
MeSH Terms: conditions — Common Bile Duct Diseases; Cholecystolithiasis; Cholangitis, Sclerosing; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ERCP without Fluoroscopy (Experimental): Non-fluoroscopic common bile duct stone extraction
  Interventions: Procedure: Endoscopic Retrograde Cholangioscopy by SpyGlass (ERCS)

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangioscopy by SpyGlass (ERCS) — Digital SpyGlass Cholangioscopy to facilitate common bile duct stone removal

SUMMARY:
This study aim to evaluated the effectiveness of Digital SpyGlass Cholangioscopy to facilitate common bile duct stone removal without fluoroscopy

DETAILED DESCRIPTION:
Patients This study recruited patients who suspected/confirmed CBDS from clinical manifestation, liver function tests and imaging studies. With CBD sized between 5 and 15 millimeters, which measured from transabdominal ultrasonography (US), computed tomography (CT), magnetic resonance cholangiopancreatography (MRCP) or endoscopic ultrasonography (EUS). The exclusion criteria were history of bile duct surgery, bile duct stricture, bile duct tumors, severe comorbid diseases, unstable vital signs, pregnancy, and coagulopathy. All patients were informed and wrote informed consent for the procedure.

Procedures Non-fluoroscopic CBDS removal was performed by experienced endoscopists, using standard side-viewing duodenoscope. After identified major papilla, the investigators performed bile duct cannulation with guidewire assisted technique. Successful cannulation confirmed by visualized bile aspiration. If the patients had difficult cannulation, double guidewire technique was used. After the successful bile duct cannulation, the investigators performed endoscopic standard sphincterotomy (EST). Precut sphincterotomy was not used in this study. Non fluoroscopic balloon extraction was performed. The balloon was pushed up to hilum then the investigators sweep until suspected complete CBD clearance. After that the investigators used digital SpyGlassTM to confirm the complete clearance of CBDS. If SpyGlassTM showed residual CBD stone, the investigators repeat balloon extraction. If SpyGlassTM showed complete clearance, the investigator proceed to perform final cholangiogram as reference standard for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected/confirmed CBDS
* CBD caliber 5-15 mm

Exclusion Criteria:

* History of bile duct surgery
* History of bile duct tumor
* History of bile duct stricture
* Severe comorbidity
* Unstable vital signs
* Pregnancy
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Success rate of SpyGlass assisted non-fluoroscopic common bile duct stones removal | 1 year

SECONDARY OUTCOMES:
Complication rate of SpyGlass assisted non-fluoroscopic common bile duct stones removal | 1 year

OTHER OUTCOMES:
Procedural time | 1 year

IPD SHARING:
Plan to Share IPD: No